CLINICAL TRIAL: NCT05330117
Title: Transcutaneous Electrical Nerve Stimulation Analgesia During Outpatient Operative Cystoscopy for Overactive Bladder: A Randomized Control Trial (TENSOB Study)
Brief Title: Nerve Stimulation Using a TENS to Provide Pain Relief During Surgery for Overactive Bladder
Acronym: TENSOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paula Doyle, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00005257
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Urinary Incontinence; Overactive Bladder; Pain, Acute
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Acute Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TENS (Experimental): In the active treatment group, the TENS unit will remain on up to 30 minutes (10 minutes pre-procedure, during the procedure and during the questionnaires).
  Interventions: Procedure: TENS
- Control TENS (Sham Comparator): The sham stimulation group will undergo the same procedure; however, the TENS stimulation current will be reduced to a minimal detectable level and turned off after 20 seconds.
  Interventions: Procedure: Control TENS

INTERVENTIONS:
Procedure: TENS — This device will then be used for deep transcutaneous nerve stimulation at the T10-L1 and S2-S4 levels. The device will be placed and activated 5 minutes before the procedure. and the device will remain active during the procedure and will be turned off as soon as the procedure is complete (procedure typically will take from 5-15 minutes). The TENS units have pre-program settings improving convenience, reproducibility and reliability. Study staff will be instructed to perform TENS using an "Acupuncture" mode on the provided TENS units. The amplitude will be adjusted to a comfortable sensation that does not cause pain using adhesive electrodes. One TENS unit is able to support 4 TENS electrodes. The TENS electrodes (8 cm x 5 cm) will be placed on bilateral paraspinal muscles. The intensity of the stimulation (Hz) will be adjusted to the subjective comfort of the subject.
  Arms: Active TENS
Procedure: Control TENS — This device will then be used for deep transcutaneous nerve stimulation at the T10-L1 and S2-S4 levels. The device will be placed and activated 5 minutes before the procedure. and the device will remain active during the procedure and will be turned off as soon as the procedure is complete (procedure typically will take from 5-15 minutes). The TENS units have pre-program settings improving convenience, reproducibility and reliability. Study staff will be instructed to perform TENS using an "Acupuncture" mode on the provided TENS units. The amplitude will be adjusted to a comfortable sensation that does not cause pain using adhesive electrodes. One TENS unit is able to support 4 TENS electrodes. The TENS electrodes (8 cm x 5 cm) will be placed on bilateral paraspinal muscles. The intensity of the stimulation (Hz) will be adjusted to the subjective comfort of the subject.
  Arms: Control TENS

SUMMARY:
This will be a double blind randomized control trial in men and women with urinary urge incontinence that are undergoing outpatient operative cystoscopy for Onabotulinumtoxin A chemo denervation as third line therapy for overactive bladder (OAB) or urinary urge incontinence (UUI). Subjects will be identified by the University of Rochester Urologists and Urogynecologists participating in the study who currently oversee urinary urge incontinence care. Subjects will be randomized into two groups. One group will be undergoing the cystoscopy with transcutaneous electrical nerve stimulation (TENS) for analgesia and the second group will have cystoscopy with placebo TENS.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women, Age ≥18 years
* Diagnosis of OAB/UUI,
* Scheduled to undergo intravesical Botox injections in the office
* Able to read/write English

Exclusion criteria:

* Currently undergoing Sacral Neuromodulation
* Cutaneous damage such as ulcers or broken skin on target treatment area
* Currently implanted cardiac pacemaker or defibrillator
* Pre-procedural use of opioids for pain management, less than 8 hours from last dose
* Participants with altered sensation below the umbilicus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Mean pain measured by Visual Analog Scale (VAS) | Baseline (Before procedure)
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.
Mean pain measured by Visual Analog Scale (VAS) | Approximately 2-5 minutes into the procedure
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.
Mean pain measured by Visual Analog Scale (VAS) | within 10 minutes after procedure
  The VAS for pain consists of a 100-mm-long horizontal line where 0-mm equals no pain and 100-mm equals worst possible pain.

SECONDARY OUTCOMES:
Mean pain measured by Likert scale | before procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Mean pain measured by Likert scale | Approximately 2-5 minutes into the procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Mean pain measured by Likert scale | within 10 minutes after procedure
  A discrete, 5-point verbal Likert scale including the following options: "no pain", "minimal pain", "moderate pain", "severe pain" and "worst pain possible" will be asked to patients
Number of participants with side effects | within 10 minutes after procedure
  A check list of vasovagal symptoms will be handed to the study team member to complete if the subject reports any light headedness, nausea or sweating.
Mean satisfaction with the procedure | within 10 minutes after procedure
  A 1-10 point satisfaction scale will be used where 10 indicates higher satisfaction.
Number of participants who guessed correctly whether they were given the active TENS or placebo TENS | within 10 minutes after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Aranda D, Panza J, Eigg M, Greenstein M, Li D, O'Brien J, Warren G, Doyle PJ. Analgesia Using Transcutaneous Electric Nerve Stimulation in Office Bladder Chemodenervation, a Randomized Controlled Trial. Urogynecology (Phila). 2024 May 1;30(5):498-504. doi: 10.1097/SPV.0000000000001424. Epub 2023 Nov 6. PMID 37930264